CLINICAL TRIAL: NCT06291389
Title: Effects of Intraoperative Peak Airway Pressure Changes on Postoperative Pulmonary Function After Muscle Plication in Abdominoplasty Operations: A Randomized Double-Blind Trial
Brief Title: Intraoperative Peak Airway Pressure Changes on Postoperative Pulmonary Function After Muscle Plication
Status: Recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Other Study IDs: RC.2.8.2023
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Abdominal Compartment Syndrome
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An abdominal panniculus excision procedure is known as an abdominoplasty (panniculectomy). Musculofascial plication is a crucial aspect of abdominoplasty, especially for patients with significant divarication of the recti muscles. This study aimed to evaluate the effect of intraoperative changes in peak airway pressure (PAP) after muscle plication on postoperative pulmonary function.

DETAILED DESCRIPTION:
Musculofascial plication is a crucial aspect of abdominoplasty, especially for patients with significant divarication of the recti muscles. This surgical procedure involves the removal of surplus skin and fat around the abdomen, known as panneculectomy, and the anterior abdominal wall muscles' laxity being tightened. This study aimed to elucidate the effect of intraoperative changes in PAP after muscle plication on postoperative pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* age ranged between 20 and 50 years old,
* American Society of Anesthesiologists (ASA) physical status classification I
* came for abdominoplasty operation

Exclusion Criteria:

* anemia or hemoglobin levels below 11g/dl
* bleeding problems
* cardiovascular disorders
* restrictive and obstructive respiratory disease
* abdominoplasty without plication.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: age ranged between 20 and 50 years old,- American Society of Anesthesiologists (ASA) physical status classification I and came for abdominoplasty operation
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative peak airway pressure (PAP) | 4 hours
  Intraoperative peak airway pressure (PAP) will be observed Pre-plication, Post- plication in supine position and Post- plication in semi-sitting position

SECONDARY OUTCOMES:
Duration of oxygen therapy | 1 week
  The duration of oxygen therapy will be recorded
Post operative Tidal Volume (Vt) (Measured by spirometer) | 24 hours postoperatively
  The post operative Tidal Volume (Vt) will be measured by spirometer and will be recorded
Post operative Respiratory Rate (RR) | 24 hours postoperatively
  The Post operative Respiratory Rate (RR) will be recorded
Hospital stay. | 1 week
  The Duration of hospital stay will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Kohaf, ph.d, Principal Investigator — Al-Azhar University
Locations (1):
- Neveen Kohaf, Tanta, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon resealable request from principle investigator
Supporting Information: Study Protocol, SAP